CLINICAL TRIAL: NCT02980276
Title: A Randomised Placebo Controlled Trial of the Effectiveness of Early MEtformin in Addition to Usual Care in the Reduction of Gestational Diabetes Mellitus Effects (EMERGE)
Brief Title: RCT Metformin for Reduction of Gestational Diabetes Mellitus Effects
Acronym: EMERGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Health Research Board, Ireland (Other); HRB Clinical Research Facility Galway (Other); University College Hospital Galway (Other); Portiuncula University Hospital (Unknown); University Hospital of Limerick (Other); University Maternity Hospital Limerick (Unknown); Clinical Research Support Unit, University of Limerick (Unknown)
Responsible Party: Principal Investigator, Fidelma Dunne, Prof. Fidelma Dunne, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NUIG-2016-01
Record Dates: First submitted 2016-11-09; First posted 2016-12-02 (Estimated); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Gestational Diabetes
Keywords: Gestational Diabetes; Diabetes; Pregnancy
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Participants randomised to the treatment arm will receive active metformin in addition to standard care. Metformin tablets will be titrated according to a dosing schedule to achieve the pre-specified glucose targets. Tablets will be in 500mg doses and will commence at 1 tablet per day (500mg) increasing to a maximum of 5 tablets per day (2500mg).
  Interventions: Drug: Metformin Hydrochloride
- Control (Placebo Comparator): Participants randomised to the placebo arm will receive placebo in addition to standard care. Placebo will be titrated according to the dosing schedule to achieve the pre-specified glucose targets. Placebo tablets will commence at 1 tablet per day and will be increased to a maximum of 5 tablets per day over 10 days as with the treatment group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin Hydrochloride — Women randomised to the metformin group will receive metformin 500mg once daily, with the dose titrated upwards every 2 days over 10 days increasing to a maximum of 2500mg Metformin daily (5 tablets) or maximum tolerated dose, in addition to usual care (exercise and MNT), and taken until delivery.
  Arms: Treatment
Other: Placebo — Women randomised to the placebo group will receive 1 placebo tablet once daily, with the dose titrated upwards every 2 days over 10 days increasing to a maximum of five placebo tablets daily, in addition to usual care (exercise and MNT), and taken until delivery.
  Arms: Control

SUMMARY:
The overall objective of the EMERGE trial is to determine whether metformin + usual care, compared to placebo + usual care (introduced at the time of initial diagnosis of GDM), reduces a) the need for insulin use, or hyperglycemia (primary outcome measure); b) excessive maternal weight gain; c) maternal and neonatal morbidities and, d) cost of treatment for women with Gestational Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Participants aged 18-50
3. Pregnancy gestation up to 28 weeks (+ 6 days) confirmed by positive pregnancy test
4. Singleton pregnancy as determined by scan
5. Positive diagnosis of Gestational Diabetes Mellitus on a Oral Glucose Tolerance Test (OGTT) according to the International Association of the Diabetes and Pregnancy Study Groups (IADPSG) criteria if any one of the following are achieved: i) Fasting glucose >/= 5.1mmol/l and <7mmol/l, or ii) 1 hour post glucose load of >/=10mmol/l, or iii) 2 hour post glucose load of >/=8.5 mmol/l and <11.1mmo/l
6. Resident in the locality and intending to deliver within the trial site

Exclusion Criteria:

1. Participants who have an established diagnosis of diabetes (Type 1, Type 2, Monogenic or secondary)
2. Participants with a fasting glucose > 7mmol/l or a 2h value > 11.1 mmol/l
3. Multiple pregnancies (twins, triplets etc.) as determined by scan
4. Known intolerance to metformin
5. Known contraindication to the use of metformin which include: i) renal insufficiency (defined as serum creatinine of greater than 130 µmol/L or creatinine clearance <60 ml/min), ii) moderate to severe liver dysfunction (aspartate aminotransferase (AST) and alanine aminotransferase (ALT) greater than 3 times the upper limit of normal, iii) shock or sepsis, and iv) previous hypersensitivity to metformin
6. Major congenital malformations or an abnormally deemed unsuitable for metformin by the site PI or attending consultant
7. Known small for gestational age (Small for gestational age (SGA) refers to foetal growth less than the 10th percentile (RCOG, 2014), or if foetal growth is deemed unsatisfactory by the treating obstetrician)
8. Known gestational hypertension or pre-eclampsia or ruptured membranes
9. Participants who have a history of drug or alcohol use that, in the opinion of the investigator, would interfere with adherence to study requirements
10. Participants with significant gastrointestinal problems such as severe vomiting, Crohn's disease or colitis which will inadvertently affect absorption of the study drug
11. Participants with congestive heart failure or history of congestive heart failure
12. Participants with serious mental illness which would affect adherence to study medication or compliance with study protocol in the opinion of the investigator
13. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 535 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Fidelma Dunne, Principal Investigator — National University of Ireland, Galway, Ireland
Locations (2):
- Ireland (2):
  - Portiuncula University Hospital, Ballinasloe, Galway
  - University Hospital Galway, Galway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dunne F, Newman C, Alvarez-Iglesias A, O'Shea P, Devane D, Gillespie P, Egan A, O'Donnell M, Smyth A. Metformin and small for gestational age babies: findings of a randomised placebo-controlled clinical trial of metformin in gestational diabetes (EMERGE). Diabetologia. 2024 Dec;67(12):2660-2666. doi: 10.1007/s00125-024-06252-y. Epub 2024 Aug 31. PMID 39215812
- [Derived] Dunne F, Newman C, Alvarez-Iglesias A, Ferguson J, Smyth A, Browne M, O'Shea P, Devane D, Gillespie P, Bogdanet D, Kgosidialwa O, Egan A, Finn Y, Gaffney G, Khattak A, O'Keeffe D, Liew A, O'Donnell M. Early Metformin in Gestational Diabetes: A Randomized Clinical Trial. JAMA. 2023 Oct 24;330(16):1547-1556. doi: 10.1001/jama.2023.19869. PMID 37786390
- [Derived] Dunne F, Newman C, Devane D, Smyth A, Alvarez-Iglesias A, Gillespie P, Browne M, O'Donnell M. A randomised placebo-controlled trial of the effectiveness of early metformin in addition to usual care in the reduction of gestational diabetes mellitus effects (EMERGE): study protocol. Trials. 2022 Sep 21;23(1):795. doi: 10.1186/s13063-022-06694-y. PMID 36131291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between June 2017 and September 2022. A total of 535 participants were randomised into the study, 502 at Galway University Hospital GUH and 33 at Portiuncula University Hospital PUH (the second site, PUH, did not start recruiting participants until February 2019).
Period: Overall Study
Arm/Group | Treatment | Control
Started | 268 | 267
Included in Analysis of Primary Outcome (262 participated in study until delivery. 264 participants included in analysis of primary outcome) | 264 | 262
Completed (Completed all study visits.) | 235 | 240
Not Completed | 33 | 27
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 18 | 18
Not completed — Death | 1 | 0
Not completed — Miscellaneous other | 10 | 4

BASELINE CHARACTERISTICS:
Population: Participants at randomisation.
Groups:
- Treatment: Participants randomised to the treatment arm received active metformin in addition to standard care. Metformin tablets will be titrated according to a dosing schedule to achieve the pre-specified glucose targets. Tablets will be in 500mg doses and will commence at 1 tablet per day (500mg) increasing to a maximum of 5 tablets per day (2500mg).
- Control: Participants randomised to the placebo arm received placebo in addition to standard care. Placebo will be titrated according to the dosing schedule to achieve the pre-specified glucose targets. Placebo tablets will commence at 1 tablet per day and will be increased to a maximum of 5 tablets per day over 10 days as with the treatment group.
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 268 | 267 | 535
Age, Categorical [Count of Participants; unit: Participants] — Age range in years at time of randomisation.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 268 | 267 | 535
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (4.9) | 34.3 (4.7) | 34.3 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 268 | 267 | 535
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African/Black | 7 | 6 | 13
  Asian | 17 | 29 | 46
  Irish Traveller | 11 | 2 | 13
  White | 219 | 209 | 428
  Other | 14 | 21 | 35
Region of Enrollment [Number; unit: Pregnancies]
  Ireland | 268 | 267 | 535
BMI [Mean (Standard Deviation); unit: kg per metre squared] — Body Mass Index in kg/meter-squared.
  kg per metre squared | 31.2 (7) | 32.1 (6.9) | 31.7 (7.1)
BMI Category >=30 [Count of Participants; unit: Participants] | 160 | 164 | 324
BMI <30 [Count of Participants; unit: Participants] | 108 | 103 | 211
Medical Card [Count of Participants; unit: Participants] | 63 | 63 | 126
Private Health Insurance [Count of Participants; unit: Participants] | 126 | 116 | 242
Unemployed [Count of Participants; unit: Participants] | 19 | 27 | 46
Current Smoker [Count of Participants; unit: Participants] | 34 | 17 | 51
History of Hypertension [Count of Participants; unit: Participants] | 12 | 4 | 16
Nulliparous [Count of Participants; unit: Participants] | 84 | 84 | 168
History of Macrosomia [Count of Participants; unit: Participants] | 57 | 44 | 101
Previous Cesarian Section [Count of Participants; unit: Participants] | 70 | 74 | 144
Previous Miscarriage [Count of Participants; unit: Participants] | 106 | 93 | 199
Prevous Pre-eclampsia [Count of Participants; unit: Participants] | 24 | 23 | 47
Previous Post-partum Hemorrhage [Count of Participants; unit: Participants] | 28 | 20 | 48
Previous Polyhydramnios [Count of Participants; unit: Participants] | 10 | 7 | 17
Previous Ante-partum Haemorrhage [Count of Participants; unit: Participants] | 20 | 15 | 35
Previous Stillbirth [Count of Participants; unit: Participants] | 2 | 2 | 4
Fasting glucose [Mean (Standard Deviation); unit: mmol/L] | 5.2 (0.45) | 5.2 (0.47) | 5.2 (0.46)
1hour Glucose Tolerance Test Result [Mean (Standard Deviation); unit: mmol/L] | 9.4 (1.9) | 9.7 (1.9) | 9.5 (1.9)
2hour Glucose Tolerance Test Result [Mean (Standard Deviation); unit: mmol/L] | 7.1 (1.6) | 7.1 (1.6) | 7.1 (1.6)
Gestational Age at Randomization [Median (Inter-Quartile Range); unit: weeks] | 27 [25 to 28] | 27 [25 to 28] | 27 [25 to 28]

OUTCOME MEASURES:

1. Primary Outcome: Primary Composite Outcome
Description: The primary efficacy outcome was achieved if any participant experienced:
  * Insulin initiation
  * Fasting glucose value >5.1 mmol/l at 32weeks or 38 weeks gestation.
Time Frame: Enrolment through delivery, an average of 16 weeks.
Population: Population of pregnancies followed up until delivery. 268 were randomised to Treatment Group, of whom 264 received Metformin as randomised. Two participants delivered outside the country; delivery and neonatal information was available for the remaining 262 participants. Among those randomised to Treatment Group, 264 Pregnancies were included in the Primary Outcome Analysis. All 262 patients randomised to placebo were followed until delivery and included in Primary Outome Analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 264 | 262
Participants | 150 | 167
Statistical Analysis 1: Comparison: Treatment vs Control; The primary analysis, as per sample size calculation, was a two-sample comparison of reduction in the proportion of women needing insulin between treatment and control arms using an exact test for a binomial response; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p = 0.13, Risk difference — The primary analysis, as per sample size calculation, was a two-sample comparison of reduction in the proportion of women needing insulin between treatment and control arms using an exact test for a binomial response; Risk Difference (RD) = -6.9, 95% CI 2-sided [-15.1 to 1.4] — Units are %

2. Primary Outcome: Insulation of Insulin
Description: Initiation of insulin treatment at any time up to delivery.
Time Frame: Enrolment through delivery, an average of 16 weeks.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 264 | 262
Participants | 101 | 134
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p = 0.004, Risk difference; Risk Difference (RD) = -12.7, 95% CI 2-sided [-21.2 to -4.3] — Units are %

3. Secondary Outcome: Time to Insulin Initiation
Description: Time to Insulin Initiation, from date of randomization until the date of delivery.
Time Frame: Time to Insulin Initiation, from date of randomization until the date of delivery, an average of 16 weeks..
Population: Pregnancies followed up until delivery.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
days | 68 (38.1) | 58.7 (37)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.001, Log Rank; Median survival times could not be calculated; time to insulin initiation would be censored at delivery in >50% of participants in treatment group

4. Secondary Outcome: Insulin Initiated
Description: Whether or not insulin was initiated at any time during the study.
Time Frame: Enrolment through delivery, an average of 16 weeks.
Population: Population of pregnancies followed up until delivery. 268 were randomised to Treatment Group, of whom 264 received Metformin as randomised. Two participants delivered outside the country; delivery and neonatal information was available for the remaining 262 participants. Among those randomised to Treatment Group, 264 Pregnancies were included in the Primary Outcome Analysis. Data for this outcome available for 263 in Treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 263 | 262
Participants | 94 | 106
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.005, Regression, Logistic; Unadjusted; Odds Ratio, log = 0.61, 95% CI 2-sided [0.43 to 0.86] — Unadjusted
Statistical Analysis 2: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.003, Regression, Logistic; Adjusted; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.38 to 0.82] — Adjusted

5. Secondary Outcome: Fasting Hyperglycemia
Description: Number of women with fasting hyperglycemia at 32wks or at 38wks gestation.
Time Frame: Measured at 32 and 38 weeks' gestation.
Population: Participants having fasting glucose levels measured at 32 and/or 38 weeks' gestation. Data available for 255 in the Treatment group and 248 in the Control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 255 | 248
Participants | 94 | 106
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.178, Regression, Logistic; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.55 to 1.12] — Unadjusted
Statistical Analysis 2: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.105, Regression, Logistic — Two-sided test comparing observed odds ratio to 1; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.48 to 1.07] — Adjusted

6. Secondary Outcome: Insulin Dose Required
Description: Insulin dose required in any participant requiring insulin.
Time Frame: Enrolment through delivery, an average of 16 weeks.
Population: Population of pregnancies followed up until delivery. 268 were randomised to Treatment Group, of whom 264 received Metformin as randomised. Two participants delivered outside the country; delivery and neonatal information was available for the remaining 262 participants. Among those randomised to Treatment Group, 264 Pregnancies were included in the Primary Outcome Analysis which includes Insulin Initiation (yes/no).
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Treatment | Control
Number analyzed (Participants) | 264 | 262
IU | 20.4 (19.8) | 2.2 (22.8)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed mean difference to zero; p = 0.17, t-test, 2 sided; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-9.3 to 1.7]

7. Secondary Outcome: Gestational Weight Gain
Description: Change in weight (kg) from randomization until last visit before delivery
Time Frame: Enrolment through delivery, an average of 16 weeks.
Population: Population of pregnancies followed up until delivery. 268 were randomised to Treatment Group, of whom 264 received Metformin as randomised. Two participants delivered outside the country; delivery and neonatal information was available for the remaining 262 participants.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
kg | 0.88 (3.31) | 1.96 (3.53)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed mean difference ratio to zero; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-1.99 to -0.42]

8. Secondary Outcome: Postpartum Impaired Fasting Glucose
Description: Impaired fasting glucose at 12 weeks postpartum
Time Frame: 12 weeks post-partum
Population: Participants followed until 12 weeks postpartum who contributed samples for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 230 | 235
Participants | 51 | 52
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.99, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.65 to 1.55]

9. Secondary Outcome: Postpartum Impaired Glucose Tolerance
Time Frame: 12 weeks postpartum
Population: Participants followed until 12 weeks postpartum who contributed samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 229 | 235
Participants | 15 | 16
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.911, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.46 to 2]

10. Secondary Outcome: Postpartum Metabolic Syndrome
Time Frame: 12 weeks postpartum
Population: Participants followed until 12 weeks postpartum who contributed samples
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 222 | 231
Participants | 20 | 25
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.519, Regression, Logistic; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.44 to 1.51]

11. Secondary Outcome: Gestational Age at Delivery
Time Frame: At delivery, an average of 16 weeks after enrolment
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
weeks | 39.1 (1.5) | 39.1 (1.6)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed mean difference to zero; p = 0.66, t-test, 2 sided; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.3 to 0.2]

12. Secondary Outcome: Mode of Delivery - Cesarian Delivery
Description: Delivered by Cesarian section.
Time Frame: At delivery, an average of 16 weeks after enrolment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
Participants | 114 | 100
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.367, Regression, Logistic; Unadjusted; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.8 to 1.85] — Unadjusted
Statistical Analysis 2: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.359, Regression, Logistic; Adjusted; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.8 to 1.87] — Adjusted

13. Secondary Outcome: Mode of Delivery - Emergency Cesarian Section
Description: Among those having cesarian section, count of emergency procedures.
Time Frame: At delivery, an average of 16 weeks after randomization.
Population: Among those having cesarian section, count of emergency procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 114 | 100
Participants | 53 | 53
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p = 1.0, Risk difference; Risk Difference (RD) = -6.5, 95% CI 2-sided [-13.9 to 12.9] — Units are %

14. Secondary Outcome: Mode of Delivery - Induced
Description: Labor induced.
Time Frame: At time of labor, an average of 16 weeks after enrolment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 259 | 262
Participants | 73 | 87
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.603, Regression, Logistic; Unadjusted; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.56 to 1.39] — Unadjusted
Statistical Analysis 2: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.621, Regression, Logistic; Adjusted; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.57 to 1.4] — Adjusted

15. Secondary Outcome: Maternal Morbidity - Pregnancy-induced Hypertension
Time Frame: From enrolment through 6 weeks postpartum, an average of 22 weeks.
Population: Participants followed from randomisation through to 12 weeks postpartum. 268 participants were randomised to Treatment Group; 264 received Metformin as randomised. Two of those participants delivered outside the country; delivery and neonatal information was available for the remaining 262 participants. 267 were randomised to Placebo, of which 262 received Placebo as randomised and were followed through to delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
Participants | 31 | 28
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.739, Regression, Logistic; Unadjusted; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.45 to 1.76] — Unadjusted
Statistical Analysis 2: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.812, Regression, Logistic; Adjusted; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.46 to 1.84] — Adjusted

16. Secondary Outcome: Maternal Morbidity - Pre-eclampsia
Description: Pre-eclampsia diagnosed during study participation
Time Frame: Enrolment through 6 weeks postpartum, an average of 22 weeks.
Population: Participants followed from randomisation through delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
Participants | 10 | 5
Statistical Analysis 1: Comparison: Treatment vs Control; Unadjusted; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.282, Regression, Logistic; Unadjusted; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.63 to 6.04] — Unadjusted
Statistical Analysis 2: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.196, Regression, Logistic; Odds Ratio (OR) = 2.14, 95% CI 2-sided [0.7 to 7.38] — Adjusted

17. Secondary Outcome: Maternal Morbidity - Antepartum Hemorrhage
Description: Any vaginal bleeding prior to delivery
Time Frame: From enrolment through delivery, an average of 16 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
Participants | 15 | 27
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.058, Regression, Logistic; Unadjusted; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.27 to 1.01]
Statistical Analysis 2: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed odds ratio to 1; p = 0.061, Regression, Logistic; Adjusted; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.27 to 1.02]

18. Secondary Outcome: Maternal Morbidity - Postpartum Hemorrhage
Time Frame: From delivery through 6 weeks postpartum.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
Participants | 51 | 63
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p = 0.24, Risk difference; Risk Difference (RD) = -4.5, 95% CI 2-sided [-11.6 to 2.5] — Units are %
Statistical Analysis 2: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p = 0.24, Regression, Logistic; Risk Difference (RD) = 0.81, 95% CI 2-sided [0.59 to 1.12] — Units are %

19. Secondary Outcome: Birthweight
Time Frame: At birth
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
grams | 3393 (527) | 3505 (510)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Regression model that adjusts for the infant's sex and maternal height and weight at randomization; p = 0.005, Regression, Linear; P value was derived from a statistical model that adjusts for the infant's sex and maternal height and weight at randomization; Median Difference (Final Values) = -113, 95% CI 2-sided [-201 to -24]

20. Secondary Outcome: Neonatal Head Circumference
Time Frame: At birth
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
cm | 34.7 (1.6) | 34.7 (1.8)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed mean difference to zero; p = 0.82, t-test, 2 sided; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.3 to 0.3]

21. Secondary Outcome: Neonatal Height
Description: Height in cm (crown-heel length)
Time Frame: At birth
Population: Pregnancies followed until delivery
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
cm | 51 (3.2) | 51.7 (3.2)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed mean difference to zero; p = 0.02, t-test, 2 sided; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.3 to -0.2]

22. Secondary Outcome: Neonatal Abdominal Circumference
Time Frame: At birth
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
cm | 33.4 (2.4) | 33.3 (2.8)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed mean difference to zero; p = 0.72, t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.5 to 0.7]

23. Secondary Outcome: Neonatal Ponderal Index
Description: Ponderal index is calculated as 100 x weight(grams)/(crown-heel length).
Time Frame: At birth
Measure: Mean (Standard Deviation); unit: grams/cm
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
grams/cm | 2.6 (0.4) | 2.6 (0.5)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed mean difference to zero; p = 0.68, t-test, 2 sided; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.1 to 0.1]

24. Secondary Outcome: Birth Weight >4000g
Time Frame: At birth
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
Participants | 20 | 39
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p = 0.02, Regression, Logistic; P value derived from a statistical model that adjusts for the infant's sex, gestational age at birth, and maternal height and weight at randomization; Risk Difference (RD) = -7.2, 95% CI 2-sided [-12.6 to -1.8] — P value derived from a statistical model that adjusts for the infant's sex, gestational age at birth, and maternal height and weight at randomization

25. Secondary Outcome: Birth Weight >90th Percentile
Time Frame: At birth
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
Participants | 17 | 39
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p = 0.003, Risk difference; P value derived from a statistical model that adjusts for the infant's sex and maternal height and weight at randomization; Risk Difference (RD) = -8.4, 95% CI 2-sided [-13.7 to -3.2] — Units are %

26. Secondary Outcome: Birth Weight <2500g
Time Frame: At birth
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
Participants | 16 | 9
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p = .012, Risk difference; Units are %. P value derived from model adjusting for the gestational age at birth, sex and maternal height and weight at randomization; Risk Difference (RD) = 2.7, 95% CI 2-sided [-1 to 6.3] — Units are %. P value was derived from a statistical model that adjusts for the infant's gestational age at birth, sex and maternal height and weight at randomization

27. Secondary Outcome: Birth Weight <10th Percentile
Time Frame: At birth
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
Participants | 15 | 7
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p = 0.13, Regression, Logistic — Units are %. P value was derived from a statistical model that adjusts for the infant's gestational age at birth, sex and maternal height and weight at randomization; Risk Difference (RD) = 3.0, 95% CI 2-sided [-0.4 to 6.5] — [estimate comment as in outcome 26, analysis 1]

28. Secondary Outcome: Neonatal Morbidity - Need for NICU Care
Time Frame: From birth until 6 weeks of life.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
Participants | 41 | 33
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p = 0.38, Risk difference; Risk Difference (RD) = 3.0, 95% CI 2-sided [-2.9 to 9] — Units are %

29. Secondary Outcome: Neonatal Morbidity - Preterm Birth
Description: Delivery at gestational age <37 weeks.
Time Frame: At birth
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 261 | 260
Participants | 24 | 17
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p = 0.33, Risk difference; Risk Difference (RD) = 2.8, 95% CI 2-sided [-2.0 to 7.3] — Units are %

30. Secondary Outcome: Neonatal Morbidity - Respiratory Distress Syndrome Requiring Respiratory Support
Time Frame: From birth until 6 weeks of life.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
Participants | 24 | 18
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p = 0.42, Risk difference; Risk Difference (RD) = 2.3, 95% CI 2-sided [-2.4 to 6.9] — Units are %

31. Secondary Outcome: Neonatal Morbidity - Jaundice Requiring Phototherapy
Time Frame: From birth until 6 weeks of life.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
Participants | 1 | 0
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p > 0.99, Risk difference; Risk Difference (RD) = 0.4, 95% CI 2-sided [-0.4 to 1.1] — Units are %

32. Secondary Outcome: Neonatal Morbidity - Major Congenital Anomalies
Time Frame: From birth until 6 weeks of life.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
Participants | 10 | 7
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p = 0.62, Risk difference; Risk Difference (RD) = 1.1, 95% CI 2-sided [-1.9 to 4.2] — Units are %

33. Secondary Outcome: Neonatal Morbidity - Apgar Score <7 at 5 Minutes
Description: The Apgar score comprises five components: 1) color, 2) heart rate, 3) reflexes, 4) muscle tone, and 5) respiration, each of which is given a score of 0, 1, or 2.
  (for example see: https://www.acog.org/clinical/clinical-guidance/committee-opinion/articles/2015/10/the-apgar-score#:~:text=The%20Apgar%20score%20comprises%20five,0%2C%201%2C%20or%202)
Time Frame: At 5 minutes after birth
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
Participants | 1 | 1
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p > 0.99, Risk difference; Risk Difference (RD) = 0, 95% CI 2-sided [-1 to 1] — Units are %

34. Secondary Outcome: Neonatal Morbidity - Neonatal Hypoglycemia
Description: serum glucose <2.6mmol/l on at least one occasion <60 minutes after delivery
Time Frame: First hour of life.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 262 | 262
Participants | 36 | 34
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Equivalence — Two-sided test comparing observed risk difference to zero; p = 0.9, Risk difference; Risk Difference (RD) = 0.7, 95% CI 2-sided [-5.1 to 6.6] — Units are %

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of randomisation through to 12 weeks postpartum, an average of 28 weeks.
Groups:
- Treatment - Mother: Women randomised to the metformin group received metformin 500mg once daily, with the dose titrated upwards every 2 days over 10 days increasing to a maximum of 2500mg Metformin daily (5 tablets) or maximum tolerated dose, in addition to usual care (exercise and MNT), and taken until delivery.
- Control - Mother: Women randomised to the placebo group received 1 placebo tablet once daily, with the dose titrated upwards every 2 days over 10 days increasing to a maximum of five placebo tablets daily, in addition to usual care (exercise and MNT), and taken until delivery.
- Treatment - Fetus/Neonate: Fetuses and babies born to women randomised to the metformin group who received metformin 500mg once daily, with the dose titrated upwards every 2 days over 10 days increasing to a maximum of 2500mg Metformin daily (5 tablets) or maximum tolerated dose, in addition to usual care (exercise and MNT), and taken until delivery.
- Control - Fetus/Neonate: Fetuses and babies born to women randomised to the placebo group who received 1 placebo tablet daily, with the dose titrated upwards every 2 days over 10 days increasing to a maximum of 5 placebo tabletes daily, in addition to usual care (exercise and MNT), and taken until delivery.
Arm/Group | Treatment - Mother | Control - Mother | Treatment - Fetus/Neonate | Control - Fetus/Neonate
All-Cause Mortality (participants affected / at risk) | 2/264 | 1/262 | 1/264 | 1/262
Serious Adverse Events (participants affected / at risk) | 79/264 | 72/262 | 107/264 | 123/262
Other Adverse Events (participants affected / at risk) | 225/264 | 247/262 | 157/264 | 172/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment - Mother (N=264) | Control - Mother (N=262) | Treatment - Fetus/Neonate (N=264) | Control - Fetus/Neonate (N=262)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Thymus enlargement (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia foetal (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Bradycardia neonatal (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Accessory auricle (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 21 (21) | 35 (35)
Aorta hypoplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Birth mark (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 7 (7) | 7 (7)
Chordee (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cleft lip (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cleft palate (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cleft uvula (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital acrochordon (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Congenital hydronephrosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congenital melanocytic naevus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Congenital naevus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 11 (11) | 12 (12)
Congenital pneumonia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital torticollis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Epispadias (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart disease congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Hypospadias (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Labial tie (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Naevus flammeus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (7)
Newborn persistent pulmonary hypertension (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pectus carinatum (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polydactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syndactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Trisomy 13 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trisomy 21 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Eye movement disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Optic atrophy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 5 (6) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (10) | 5 (6) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenogastric reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infantile colic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infantile vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Inadequate analgesia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholestasis of pregnancy (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy to vaccine (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 7 (8) | 6 (6)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Endometritis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Omphalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 4 (4) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Foetal exposure during delivery (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reaction to previous exposure to any vaccine (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Poor feeding infant (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infantile haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 4 (5) | 7 (8)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
False labour (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 15 (18) | 17 (17) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 7 (9) | 7 (8)
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Neonatal disorder (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Unstable foetal lie (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Uterine irritability (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decrease neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ketonuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urethral meatus stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cyanosis neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 10 (10) | 10 (10)
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 7 (7) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Antibiotic prophylaxis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Hepatitis B immunisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Subgaleal haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment - Mother (N=264) | Control - Mother (N=262) | Treatment - Fetus/Neonate (N=264) | Control - Fetus/Neonate (N=262)
Anaemia (Blood and lymphatic system disorders) | 66 (70) | 77 (79) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 5 (5) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Bradycardia foetal (Cardiac disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1)
Bradycardia neonatal (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foetal heart rate deceleration abnormality (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neonatal tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 6 (6)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 11 (11) | 14 (15) | 0 (0) | 0 (0)
Tachycardia foetal (Cardiac disorders) | 2 (2) | 4 (5) | 1 (1) | 2 (2)
Congenital acrochordon (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital skin dimples (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 6 (6) | 10 (10)
Congenital uterine anomaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 6 (6) | 7 (7)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 6 (6) | 8 (8)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 8 (8) | 11 (12)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (4)
Vision blurred (Eye disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 11 (11) | 11 (11) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 78 (82) | 23 (24) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 31 (34) | 27 (31) | 6 (6) | 6 (6)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal skin tags (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 5 (5) | 7 (7) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 10 (13) | 1 (1) | 2 (2)
Duodenogastric reflux (Gastrointestinal disorders) | 1 (1) | 5 (5) | 27 (27) | 20 (20)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 9 (9) | 2 (2) | 0 (0) | 0 (0)
Infantile colic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 7 (7) | 3 (3)
Infantile vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 5 (5)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 6 (7) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Application site vesicles (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Developmental delay (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug intolerance (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site atrophy (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Mass (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 30 (35) | 40 (45) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 5 (5) | 9 (9)
Vessel puncture site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (3) | 8 (9) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Amniotic cavity infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 8 (10)
COVID-19 (Infections and infestations) | 17 (17) | 16 (17) | 6 (6) | 2 (3)
Candida infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Endometritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (6) | 7 (7) | 2 (2) | 1 (1)
Genital herpes (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mumps (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 12 (12) | 12 (12) | 0 (0) | 2 (2)
Omphalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 11 (12) | 8 (8)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perineal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 4 (6) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Puerperal pyrexia (Infections and infestations) | 5 (5) | 13 (13) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 18 (20) | 21 (23) | 4 (4) | 9 (9)
Rhinitis (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 6 (6) | 7 (7) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 35 (42) | 46 (56) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 14 (15) | 12 (12) | 0 (0) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 6 (6) | 4 (5)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental restoration failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 5 (5) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Repetitive strain injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin pressure mark (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vascular access site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound decomposition (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amniotic fluid index decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amniotic fluid index increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amniotic fluid volume decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amniotic fluid volume increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Antimicrobial susceptibility test (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood gases abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood ketone body (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 4 (4) | 9 (10) | 0 (0) | 1 (1)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 5 (5) | 2 (2)
Chest X-ray abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dural tap (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Streptococcus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ultrasound scan abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ultrasound uterus abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 18 (23) | 19 (23) | 1 (1) | 0 (0)
Urine uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cow's milk intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Dairy intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 15 (15) | 7 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired fasting glucose (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Poor feeding infant (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Axillary mass (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 10 (10) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delayed fontanelle closure (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertonia neonatal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypotonia neonatal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Symphysiolysis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infantile haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Intracystic breast papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cluster headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 7 (9) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foetal movement disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fontanelle bulging (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 30 (35) | 38 (46) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 7 (8) | 2 (3) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Poor sucking reflex (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 7 (8) | 0 (0) | 0 (0)
Psychogenic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Sore throat (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Birth trauma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Chronic villitis of unknown etiology (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foetal growth abnormality (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2) | 1 (1) | 2 (2)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 56 (67) | 65 (79) | 2 (2) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothermia neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 42 (45) | 37 (38)
Neonatal disorder (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Placenta accreta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Placental disorder (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Placental infarction (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Poor weight gain neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shoulder dystocia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Umbilical cord abnormality (Pregnancy, puerperium and perinatal conditions) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical cord vascular disorder (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Uterine hyperstimulation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine irritability (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decrease neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 5 (5) | 9 (9)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perinatal depression (Psychiatric disorders) | 13 (13) | 9 (9) | 0 (0) | 0 (0)
Bence Jones proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Crystalluria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 13 (14) | 9 (10) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Ketonuria (Renal and urinary disorders) | 33 (38) | 27 (34) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 48 (59) | 40 (56) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureteral disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethral perforation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bartholin's cyst (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Breast engorgement (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 5 (5) | 2 (2) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast ulceration (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical cyst (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ectropion of cervix (Reproductive system and breast disorders) | 9 (9) | 3 (3) | 0 (0) | 0 (0)
Genital blister (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lactation disorder (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nipple exudate bloody (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 4 (4) | 3 (4) | 0 (0) | 0 (0)
Penile swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal erythema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Testicular retraction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Uterine malposition (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal cyst (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 15 (17) | 9 (9) | 0 (0) | 0 (0)
Vaginal haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Vulval disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 6 (6) | 3 (3) | 4 (4)
Cyanosis neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Grunting (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (6)
Nasal septum haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 6 (6)
Neonatal respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 18 (18) | 20 (20)
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acne infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Erythema ab igne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 9 (9) | 7 (7)
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polymorphic eruption of pregnancy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (10) | 16 (17) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 9 (9) | 9 (10) | 0 (0) | 0 (0)
Rash neonatal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (6) | 6 (6)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin weeping (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient neonatal pustular melanosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical haematoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Antibiotic prophylaxis (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Retained placenta operation (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tooth repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Extravasation blood (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Haematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 11 (11) | 4 (4) | 0 (0) | 0 (0)
Inferior vena cava syndrome (Vascular disorders) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Subgaleal haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 4 (5) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT02980276/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT02980276/SAP_001.pdf